CLINICAL TRIAL: NCT02205944
Title: The Impact of Exercise on Vascular Remodeling, Arteriovenous Fistula Creation and Use in Patients With Chronic Kidney Disease: A Randomized Controlled Trial
Brief Title: Impact of Presurgical Exercise on Hemodialysis Fistula Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Charmaine Lok, Professor of Medicine, University of Toronto, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAPCR-ID: 13-6763-AE
Record Dates: First submitted 2014-07-09; First posted 2014-08-01 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; hemodialysis; vascular access; arteriovenous fistula; forearm exercise
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): The control group will receive routine vascular access pre-op teaching and care.
- Normal Exercise Group (Experimental): Group 1 (Normal Exercise Group): progressive handgrip exercise
  Group 2 (Restricted Blood Flow Exercise Group): progressive handgrip exercise with controlled tourniquet
  Interventions: Other: Progressive Handgrip Exercise

INTERVENTIONS:
Other: Progressive Handgrip Exercise — Group 1 (Normal Exercise Group): Daily, at home for 20 minutes using an adjustable handgrip trainer up to 8 weeks prior to a scheduled surgery for fistula creation. The exercise intensity is tailored using the Borg CR100 scale (Borg & Borg, 2001).
  Group 2 (Restricted Blood Flow Exercise Group): Same as the exercise performed by Group 1 with controlled tourniquet.
  Arms: Normal Exercise Group

SUMMARY:
The purpose of this research study is to determine whether two different types of forearm exercise, performed before fistula creation surgery, can improve surgery success and fistula maturation.

DETAILED DESCRIPTION:
This is a randomized, double blinded controlled trial to study the impact of handgrip exercise prior to surgical creation of hemodialysis fistula on vascular remodelling and fistula maturation in chronic kidney disease patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age>18 years old) with chronic kidney disease
2. Hemodialysis is their renal replacement therapy (RRT) modality
3. Deemed eligible for an arteriovenous fistula
4. Anticipated RRT start < 3 months (from the time of vascular surgery assessment) if predialysis
5. Scheduled surgical creation of fistula aniticpated >= 8 weeks
6. Able to follow instructions for an exercise intervention
7. Able to provide informed written consent

Exclusion Criteria:

1. Life expectancy < 6 months
2. Need for urgent vascular access (i.e. <4 weeks)
3. Pre-existing fistula distal to site of newly scheduled fistula
4. Ipsilateral central stenosis or occlusions not amenable to correction
5. Contraindications or unable to perform handgrip exercise

   * Unable to withstand transiently raised systolic blood pressure (SBP) by 35 mmHg, and diastolic (DBP) by 25 mmHg
   * severe upper extremity arthritis or other pain
6. Contraindications to general exercise

   * Poorly controlled blood pressure - SBP>180, DBP>90; SBP<110, DBP<50
   * NYHC IV heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Late dialysis suitability failure | 6 months after surgery
  Late dialysis suitability failure is a fistula that, despite radiological or surgical intervention, cannot be used successfully for dialysis by the sixth month following its creation.

SECONDARY OUTCOMES:
Change of intra-access flow and vascular diameters at predetermined distances from the fistula anastomosis; arterial stiffness and endothelial function on a randomly determined sub sample of patients. | Baseline, week 9 and week 11
  Ultrasound measurements using duplex ultrasonography
Plasma cGMP (cyclic guanosine monophosphate) and NO (nitric oxide) levels | Baseline, week 9 and week 11
  cGMP and NO will be sampled in blood plasma collected immediately prior to ultrasound assessment
Fistula maturation | 6 weeks after surgery
  A fistula will be deemed mature if either criterion are met: 1) the National Kidney Foundation Disease Outcomes Quality Initiative 'rule of six' , or 2) the draining vein diameter is > 4 mm with intra-access flows > 500 ml/min AND an experienced hemodialysis nurse, blinded to group allocation, deems maturation to have occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Charmaine Lok, MD, FRCPC, MSC, Principal Investigator — University Health Network, Toronto; Chris Chan, MD, Principal Investigator — University Health Network, Toronto; Jamie Macdonald, PhD, Principal Investigator — Bangor University; David Cherney, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital - UHN, Toronto, Ontario, Canada